CLINICAL TRIAL: NCT00140179
Title: Valnoctamide as a Valproate Substitute With Low Teratogenic Potential: Double-Blind Controlled Clinical Trial
Brief Title: Valnoctamide in Mania
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Yuly Bersudsky, Ben Gurion University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMHC-3658
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Mania; Schizoaffective Disorder, Manic Type
Keywords: valnoctamide; teratogenicity; double-blind; mania
MeSH Terms: conditions — Mania; Psychotic Disorders; Teratogenesis | interventions — valnoctamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: valnoctamide

SUMMARY:
Valproic acid is a leading mood stabilizer for the treatment of bipolar disorder. Its well-known teratogenicity limits its use in young women of childbearing age. According to toxicologic studies the teratogenicity of valproate stems from its free carboxylic group. Valnoctamide is an isomer and an analog of valpromide. Unlike valpromide, valnoctamide does not undergo a biotransformation to the corresponding free acid. It is also likely or at least possible that valnoctamide is anti-bipolar. In mice valnoctamide has been shown to be distinctly less teratogenic than valproate. An injection at day 8 of gestation produced only 1% exencephaly (as compared to 0-1% in control mice and 53% in valproate treated mice).

The investigators are performing a double-blind controlled trial of valnoctamide as an anti-bipolar drug. If shown to be anti-bipolar, valnoctamide could be an important valproate substitute for young women with bipolar disorder who are at risk of pregnancy. Patients newly admitted to the Beersheva Mental Health Center may participate if they meet Diagnostic and Statistical Manual of Mental Disorders - 4th edition (DSM-IV) criteria for mania or schizoaffective disorder, manic type. Patients admitted to the study are treated with risperidone at doses of the physicians' discretion beginning with 2 mg daily on days 1 and 2. Valnoctamide or placebo is begun at doses of 600 mg per day (200 mg three times daily) and increased to 1200 mg (400 mg three times daily) after four days.

Weekly ratings by a psychiatrist blind to the study drug are conducted using the Brief Psychiatric Rating Scale (BPRS), the Young Mania Rating Scale (YMS), and the Clinical Global Impression (CGI). Weekly blood is drawn for drug levels of valnoctamide to be measured by gas chromatography. Each patient receives valnoctamide or placebo for 5 weeks.

Low teratogenic mood stabilizers are a high priority for current research.

DETAILED DESCRIPTION:
Valproic acid is a leading mood stabilizer for the treatment of bipolar disorder. Its well-known teratogenicity limits its use in young women of childbearing age (1-3). The alternative mood stabilizers such as lithium and carbamazepine also have teratogenic potential so the treatment of bipolar disorder in young women is problematic. The difficulties are particularly acute in those young women patients who respond well to anti-bipolar therapy and maintain or begin normal interpersonal and marital relations and desire to have children.

One approach to this problem has been the search for valproic acid derivatives with less teratogenic potential (4). According to toxicologic studies the teratogenicity of valproate stems from its free carboxylic group (2, 3). Valpromide is an amide derivative of valproate without the suspect free carboxylic group. It was synthesized and marketed and has anticonvulsant efficacy, at least as good as valproic acid (1). There are some reports of its efficacy in bipolar disorder as well (5). In some animal species, only a small amount of valpromide is metabolized to valproic acid. However, in humans valpromide is metabolized to a large degree to valproic acid and so it does not solve the problem of teratogenicity (1, 6).

Valnoctamide is an isomer and an analog of valpromide. Unlike valpromide, valnoctamide does not undergo biotransformation to the corresponding free acid (6-9). In animal studies it is at least as anticonvulsant as valproate and valpromide (1, 6, 10). It has been marketed as an anxiolytic and sedative in several European countries (as Nirvanil) including Italy, Holland and Switzerland but has not actively been promoted as an anticonvulsant. It was marketed in the USA as Axiquel by McNeil in the 1970's. Unfortunately, despite considerable efforts we have not been able to obtain pharmacovigilance data from this period. Given its equivalence to valproate and valpromide as an anticonvulsant in animal models of epilepsy (1, 6, 10), it is reasonable to assume that valnoctamide is also anticonvulsant in humans. It is also likely or at least possible that valnoctamide is anti-bipolar. In mice valnoctamide has been shown to be distinctly less teratogenic than valproate (11). Injection at day 8 of gestation produced only 1percent exencephaly (as compared to 0-1percent in control mice and 53 percent in valproate treated mice). Embryolethality rates showed similar results: 52 percent with valproate vs. 5percent in the controls and 2 percent with valnoctamide.

Valnoctamide's patent is expired (12) and it is not the property of any major pharmaceutical company. Pharmaceutical company support cannot be obtained for our trial; therefore it is investigator initiated.

Valnoctamide will be synthesized for our study by Banyan Chemical in India (which has been inspected by the FDA) by GLP (good laboratory practice) in a manner acceptable for human use by the Israel Ministry of Health (and in principle for an IND by the FDA). Banyan manufactures at the same site generic compounds, atenolol for instance, sold in the USA and distributed by international companies, Novartis for instance.

Study Design:

The study has been submitted to our Helsinki Committee and only patients who give informed written consent will be accepted. Patients newly admitted to the Beersheva Mental Health Center may participate if they meet DSM-IV criteria for mania or schizoaffective disorder, manic type. Minimal Young Mania Scale = 20. Only patients admitted to the hospital within the previous 72 hours will be eligible for the study. Exclusion criteria will be as in previous studies of mania with this design by our group (15-17) and will include drug abuse, active physical illness, and of course pregnancy.

Patients admitted to the study will be treated with risperidone at doses of physicians' discretion beginning with 2 mg daily on days 1 and 2. On days 3 and 4 the risperidone dose could be increased to a maximum of 4 mg daily or decreased to 1mg daily. On days 5 to study end the dose could be increased to a maximum of 6 mg daily or decreased to a minimum of 1mg (see ref #18). Dose of risperidone will be a secondary outcome measure (see reference #15 & #16). No washout from previous medication is required but patients who received depot neuroleptics within the past 2 weeks or more than 300 mg of chlorpromazine equivalents in the past three days will be excluded. Trihexyphenidyl (up to 4 mg daily) will be available as necessary for extrapyramidal symptoms and benzodiazepines for sleep. Valnoctamide or placebo will be begun at doses of 600 mg per day (200 mg three times daily) and increased to 1200 mg (400 mg three times daily) after four days. This dose is based on relative anticonvulsant effects of valproate and valnoctamide in animal studies (1, 6, 10).

Patients will receive valnoctamide or identical capsules of placebo as assigned by the control psychiatrist according to random order; manic and schizoaffective manic patients will be randomized separately. Weekly ratings by a psychiatrist blind to the study drug will be conducted using the Brief Psychiatric Rating Scale (BPRS), the Young Mania Rating Scale (YMS), and the Clinical Global Impression (CGI). Primary outcome measure will be BPRS. Weekly blood will be drawn for drug levels of valnoctamide to be measured by gas chromatography (19). Each patient will receive valnoctamide or placebo for 5 weeks.

Power Analysis:

We have demonstrated significant effects as add-on in mania in this design with lithium (15), carbamazepine (16), and phenytoin (17). Each study had an N of about 40 patients, recruited over 18 months in each study. In each study as in the present proposal, a mood stabilizer or potential mood stabilizer was added to haloperidol at doses of physician's discretion for five weeks.

Lithium adds clinically and statistically significant benefit to haloperidol treatment of mania (15) as does carbamazepine (16) and phenytoin (17). Such an "add-on" design is consistent with clinical practice and makes sense since dopamine blockers and mood stabilizers probably work by different mechanisms in mania. Valproate is typically used clinically in acute mania as an add-on to neuroleptics as well. Three positive studies published in excellent journals (15-17) from our group using this design are probably better than formal power analysis, which depends on a range of assumptions that are collapsible into the experience of our three studies. Because the prior probability of an effect of valnoctamide is lower than that of the above well-known compounds, we suggest recruitment of 80 patients over 36 months to adequately power this study rather than the 40 patients in each of our previous studies. Since valnoctamide is no longer patented, orphan drug procedures or a use patent of the type granted to Abbott for divalproex sodium will be necessary to make this drug available for bipolar patients at risk for pregnancy in the future. An adequately powered study is therefore important at this stage.

References

1. Bialer M, Haj-Yehia A, Badir K, Hadad S: Can we develop improved derivatives of valproic acid? Pharm World Sci 1994; 16(1):2-6.
2. Nau H, Headrick X: Valproic acid teratogenesis. ISI Atlas Sci Pharmacol 1987; 1:52-56
3. Nau H, Hauck RS, Ehlers K: Valproic acid-induced neural tube defects in mouse and human: aspects of chirality, alternative drug development, pharmacokinetics and possible mechanisms. Pharmacol Toxicol 1991; 69(5):310-21.
4. Bialer M: Pharmacokinetic considerations in the design of better and safer new antiepileptic drugs. J Control Release 1999; 62(1-2):187-92.
5. Lemoine P, Fondarai J, Faivre T: Valpromide increases amplitude of heart rate circadian rhythm in remitted bipolar and unipolar disorders. A placebo-controlled study. Eur Psychiatry 2000; 15(7):424-32.
6. Bialer M: Clinical pharmacology of valpromide. Clin Pharmacokinet 1991; 20(2):114-22.
7. Bialer M, Haj-Yehia A, Barzaghi N, Pisani F, Perucca E: Pharmacokinetics of a valpromide isomer, valnoctamide, in healthy subjects. Eur J Clin Pharmacol 1990; 38(3):289-91.
8. Haj-Yehia A, Bialer M: Pharmacokinetics of valpromide isomer valnoctamide in dogs. J Pharm Sci 1988; 77:831-834.
9. Pisani F, Haj-Yehia A, Fazio A, Artesi C, Oteri G, Perucca E, Kroetz DL, Levy RH, Bialer M: Carbamazepine-valnoctamide interaction in epileptic patients: in vitro/in vivo correlation. Epilepsia 1993; 34(5):954-9.
10. Loscher W, Nau H: Pharmacological evaluation of various metabolites and analogues of valproic acid. Anticonvulsant and toxic potencies in mice. Neuropharmacology 1985; 24(5):427-35.
11. Radatz M, Ehlers K, Yagen B, Bialer M, Nau H: Valnoctamide, valpromide and valnoctic acid are much less teratogenic in mice than valproic acid. Epilepsy Res 1998; 30(1):41-8.
12. US Patent 3,056,726 (1962): alpha-ethyl-beta-methylvaleramide for mental hyperirritability. McNeil Laboratories Inc.
13. Phiel CJ, Zhang F, Huang EY, Guenther MG, Lazar MA, Klein PS: Histone deacetylase is a direct target of valproic acid, a potent anticonvulsant, mood stabilizer, and teratogen. J Biol Chem 2001; 276(39):36734-41.
14. Shaltiel G, Shamir A, Belmaker RH, Greenberg ML, Agam G: Valproate inhibits inositol-P synthase: mood stabilization by inositol depletion elaborated. submitted
15. Biederman J, Lerner Y, Belmaker RH: Combination of lithium carbonate and haloperidol in schizo-affective disorder: a controlled study. Arch Gen Psychiatry 1979; 36(3):327-33.
16. Klein E, Bental E, Lerer B, Belmaker RH: Carbamazepine and haloperidol v placebo and haloperidol in excited psychoses. A controlled study. Arch Gen Psychiatry 1984; 41(2):165-70.
17. Mishory A, Yaroslavsky Y, Bersudsky Y, Belmaker RH: Phenytoin as an antimanic anticonvulsant: a controlled study. Am J Psychiatry 2000; 157(3):463-5.
18. Yatham LN, Grossman F, Augustyns I, Vieta E, Ravindran A: Mood stabilisers plus risperidone or placebo in the treatment of acute mania. International, double-blind, randomised controlled trial. Br J Psychiatry 2003; 182:141-7.
19. Bialer M, Hoch B: Rapid gas chromatographic assay for monitoring valnoctamide in plasma. J Chromatogr 1985; 337:408-411.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60
* Males or females
* DSM-IV criteria for mania or schizoaffective disorder, manic type
* Minimal Young Mania Scale = 20
* Admittance to hospital within previous 72 hours

Exclusion Criteria:

* Any active physical illness
* Pregnancy
* Drug or alcohol abuse
* Suicidal or violent ideation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2004-09; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale
Young Mania Rating Scale
Clinical Global Impression

CONTACTS AND LOCATIONS:
Overall Officials: RH Belmaker, MD, Study Director — Ben Gurion University of the Negev + Beersheva Mental Health Center
Locations (3):
- Israel (3):
  - Hemek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Beersheva Mental Health Center, Beersheva